CLINICAL TRIAL: NCT06206551
Title: Implementing Spiritual Care in Inpatient Palliative Care
Acronym: SCPC
Status: Completed | Type: Observational
Sponsor: University Hospital Muenster (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-465-b-S
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-11

CONDITIONS: Cancer; Heart Failure; Chronic Obstructive Pulmonary Disease; Lateral Sclerosis
MeSH Terms: conditions — Neoplasms; Heart Failure; Pulmonary Disease, Chronic Obstructive; Motor Neuron Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prospective patients: Patients who are on the palliative care ward or who are being treated by the palliative consultation service at the University Hospital Muenster.
  Interventions: Other: Spiritual Needs Questionnaire
- Restrospective patients: Patients who were on the palliative care ward or were treated by the palliative consultation service at University Hospital Muenster during the same period in the previous year.

INTERVENTIONS:
Other: Spiritual Needs Questionnaire — This questionnaire captures the spiritual needs of patients and is used in its short version (screener).This questionnaire is used as part of standard treatment for all palliative care inpatients.
  Groups: Prospective patients

SUMMARY:
The goal of this observational study is to is to ascertain the spiritual needs of palliative patients in a standardized manner using the Spiritual Needs Questionnaire and to promptly address those needs by (specialized) spiritual care.

To determine whether the effort of implementing the Spiritual Needs Questionnaire on a sustainable basis on the one hand brings the expected benefit to the patients and on the other hand can be provided by the pastoral care personnel, at Muenster University Hospital (specialized) spiritual care interventions will be documented in detail and retrospectively and prospectively collected data will be compared.

ELIGIBILITY:
Inclusion Criteria:

* All individual indication for general and specialised Palliative Care in clinical setting/routine (e.g.):

  * Progressive, malign tumours
  * Progressive, chronic obstructive pulmonary disease
  * Patients with progressive disease and limited life expectancy (< ca. 12 months)
* Patients attended by Palliative Caregivers in counselling services or on palliative ward
* Life expectancy > 2 weeks
* Sufficient comprehension of German language and writing that allows an autonomous or supported completion of the questionnaire.
* Existence of an independently signed written consent.

Exclusion Criteria:

* Severe cognitive impairment
* capacity for consent lacking or impaired
* impaired comprehension of German language and writing that would not allow an autonomous or supported completion of the questionnaire.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients assigned to general and specialized Palliative Care due to justifying indications like progressive malign and non-malign diseases that need inpatient treatment provided by either counselling services or on palliative ward.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of standardized and evidence-based recordation and implementation of Spiritual Care in Palliative Care | 6 months
  Feasibility of standardized and evidence-based recordation and implementation of Spiritual Care in Palliative Care based on the number of interventions provided by general and/or specialized Spiritual Care for patients with ascertained needs detected by the validated Spiritual Needs Questionnaire in German language.

SECONDARY OUTCOMES:
Recordation of needs for general / specialized spiritual care in palliative care | 6 months
  Recordation of needs for general / specialized spiritual care in palliative care consultation service and palliative ward of a university tertiary care hospital.
Differences in use and outcomes comparing standardised and non-standardised evaluation of spiritual care needs (comparison with retrospective data). | 6 months
  s. title
Examination of further descriptive and analysing comparisons of retrospective data and intervention group. | 6 months
  s. title

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Lenz, Prof. Dr. med., Principal Investigator — University Hospital Muenster
Locations (1):
- University Hospital Muenster, Münster, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No